CLINICAL TRIAL: NCT04290650
Title: The AkuSleep Study- Treating Sleep Disturbances in Patients With Psychotic Symptoms in an Acute Ward Setting Using Cognitive Behavioral Treatment Techniques
Brief Title: Sleep Disturbances in Patients With Psychotic Symptoms (AkuSleep)
Acronym: AkuSleep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Ingrid Dieset, MD, PhD, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50984
Record Dates: First submitted 2020-02-24; First posted 2020-03-02 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Sleep Disturbance; Psychotic Disorders
Keywords: Sleep Disturbance; Psychotic Disorders
MeSH Terms: conditions — Parasomnias; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified CBT for insomnia (Other): All patients admitted to one of the psychosis ward will be offered the same customized treatment focusing on sleep in addition to treatment as usual.
  Interventions: Behavioral: Modified CBT for insomnia
- Treatment as usual (Other): All patients admitted to the other two psychosis wards will only receive treatment as usual.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Modified CBT for insomnia — Nurses who are working closely with the patients around the clock will perform an adjusted and modified version of CBT for sleep disturbances, in addition to standard evidence based treatment for psychosis and affective disorders as per today.
  Arms: Modified CBT for insomnia
Behavioral: Treatment as usual — All patients on the two other psychosis wards will receive standard evidence based treatment for psychosis and affective disorders as per today.
  Arms: Treatment as usual

SUMMARY:
Sleep disturbance is recognized as a major problem for patients with psychosis and is seen in nearly all patients admitted in acute crisis to a psychiatric hospital.

Cognitive behavioral treatment is recommended as first-line treatment for insomnia in national and international guidelines. This study explores effect of adapting the milieu therapy to comply with the principles of CBT for insomnia. Our aim is to rethink our day to day psychological interventions and our around the clock milieu therapy for patients with acute and severe mental illness in light of established knowledge on how sleep is obtained and maintained.

DETAILED DESCRIPTION:
Sleep disturbances are highly prevalent among patients admitted to any hospital ward, but in particular in psychiatric patients where insomnia and poor sleep quality is a major clinical challenge.

Approximately 950 patients are admitted to The Acute Psychiatric Department at Oslo University each year. The majority of the patients (approximately 450) admitted for more than 48 hours have a severe psychotic disorder and after being evaluated by a psychiatrist upon admittance, they are allocated to one of three similar wards specialized in the treatment of psychosis. A majority of the patients experience sleep difficulties both in terms of insomnia and problems regulating circadian rhythm. Psychiatric wards in general offer several challenges to sleep, including limited access to natural daylight, noisy environment and frequent observations by staff during night for risk management purposes. A part from offering medication which the patient often declines, staff members possess little means as to how to cope with noise and agitation at night time due to frustrated patients unable to find rest.

In September 2019 our department started organizing the treatment for psychotic patients in three similar wards ("psychosis wards") and patients were allocated to a ward according to their date of birth. Nurses are stationed permanently at each ward, while psychiatrist and psychologists make up a "specialist pool" serving all three psychosis wards. One of the main intentions for organizing the department and treatment this way is to ensure that all patients with psychotic disorders receive the same treatment according to recommended guidelines.

The aim of our study is to rethink our day to day psychological interventions and our around the clock milieu therapy for our patients with acute and severe mental illness in light of established knowledge on how sleep is obtained and maintained. After making physical adjustments to the ward environment and training allocated nurses in modified CBT techniques, the AkuSleep intervention will start up in March 2020 and will be carried out for up to six months. All patients admitted one of the psychosis wards will be offered the same customized treatment focusing on sleep, whereas all the patients admitted to the other two psychosis wards will receive treatment as usual (TAU). Upon discharge, all patients admitted to the Department of Acute Psychiatry who are able to give informed consent are asked to give a broad consent allowing us to systemize clinical information from hospital records for research purposes.

The AkuSleep protocol is as follows:

1. Identify the nature of the patient's sleeping problems and discuss suitable adjustments with the patient. These adjustments would typically be to focus on circadian rhythm, such as getting up in the morning at set times, avoiding coffee and strenuous physical and emotional activities at night time, avoiding staying in bed when sleep is not achieved and optimizing light/dark exposure. An acute ward setting such as ours is often noisy and many of our patients have restrictions due to security reasons which limit the access to natural day light. Simple physical measures will be implemented such as providing ear plugs, providing night lamps so that staff don't need to turn on lights on rounds, secure speakers so that the patients may listen to soothing music, easy blinds to secure a dark room at night and bean bags (or chairs) in every room so that the patient can get out of bed when sleep is not achieved. The use of daylight lamps will be offered for patients who due to security reasons or otherwise are denied access to natural daylight.
2. Trained nurses will perform a short 20 minute daily session with the patient addressing tailored measures in accordance with the modified CBT for insomnia. Assessment of the individual patient's specific sleeping problems is vital for an effective treatment. Sleeping problems/disorders typically falls in to three categories; disturbance in the sleep/wake homeostasis, disturbance in the circadian rhythm and/or hyperarousal. Detecting the nature of the sleeping disorder, maintenance factors and individual goals for treatment will give way to a sleep-focused case formulation that will guide further strategies. The use of sleep and activity monitoring devices will be offered for those who find it useful. Information from monitoring devices will be used for the purpose psychoeducation and as basis for the sleep diary and relevant information will be registered in the clinical records. Data from monitoring devices will not be stored electronically. Intentions available for the patient and therapist are gathered from CBT for insomnia and will involve establishing a firm associations between bed and sleep through the use of stimulus control and the setting of a consistent sleep window (time spent in bed); activity scheduling to promote good wake-up routines and help build up necessary sleep pressure; targeting hyperarousal through systematic wind-down strategies, relaxation training etc. Psychotic symptoms such as hallucinations and delusions are also prone to give disturbance in the ability to either getting to or staying asleep. These symptoms will be incorporated in the specific formulation for treatment and management of the symptoms will be a part of later strategies promoting good sleep hygiene. The implemented measures will be monitored and evaluated throughout the whole period so that adjustments can be made on a daily basis and in accordance with the formulation and the patient's goals. The details of the individual treatment progress will be written in a patient owned workbook, giving all trained staff members an opportunity to step in at any time to continue the therapeutic work. The workbook will be given to the patient at their time of discharge with instructions of further use.

The teaching of the nursing staff will cover topics to enable them to give psychoeducation about the function and the architecture of sleep, to assess sleep quality and disturbance and to create a case formulation. Nursing staff will be trained in specific cognitive techniques that target night time worries and the handling of hallucinations/voices. The interventions will be manualized, securing equality in treatment for all patients. A clinical psychologist with CBT training, stationed at the ward, will take part in the initial assessment and will offer support in the creating the case formulation. The standardized evaluation using symptom checklists and sleep checklists will also be conducted by the psychologist or doctor in charge. Supervision will be given in groups led by a clinical psychologist on a weekly basis as well as ad hoc troubleshooting and problem solving on a daily basis. The individual treatment will include an activity plan for each patient prepared in close collaboration with our wards occupational therapist concerning. This will involve good wake up routines and winding down-routines, light exposure to reestablish circadian rhythm and activating activities to counteract the need for daytime naps that disturbs the build-up of sleep pressure. Much of the described measures are already part our established inpatient nursing services or "treatment as usual". The focus of our project, however, will be to systemize these interventions in light of a 24 hour cycle aimed specifically to target the promotion of good sleep. Before discharge, the psychologist or doctor in charge will conduct a reevaluation using symptom checklist as well as an interview focusing on lessons learned and tool acquired by our patients struggling with chronic sleep disturbances in how to cope with these challenges after their discharge.

All patients on all three psychosis wards will receive standard evidence based treatment for psychosis and affective disorders as per today. All patients on the two wards not receiving the treatment protocol will also be offered to wear a monitoring device on order to register potential sleep disturbances. All patients who choose to wear a monitoring device, will be offered a psychoeducative session with a psychologist trained in CBT upon discharge.

Primary outcome will be the quantity and quality of sleep as measured by clinical records on sleep duration, sleep onset, number of awakenings, bed time, rise time and medication used. Secondary outcomes will be symptom load as measured by clinical records of nursing category (PK) and Brøset Violence Checklist (BVC), symptom measurements for psychosis (PANSS), for mania (YMRS) and global assessment of function (GAF). In addition daily dosage of medication such as antipsychotics, mood stabilizers, benzodiazepines and sleep inducing medication, as well as registered aggressive events will be measured. In most cases the patient is admitted involuntary and time until their legal status is changed from involuntary to voluntary will be calculated as a measurement of insight and health improvement. Finally, average number of bed days, ward level of violence and wards cost of medication for the three wards will be calculated and compared for all patients admitted during the study period.

Patients admitted to an acute psychiatric ward are very often not able to give informed consent upon admittance due to psychotic symptoms. Those who are able to give informed consent upon discharge will be asked to sign a broad consent. For those patients who consent upon discharge, data will be gathered for all patients on all three psychosis wards and compared against each other. Aggregated and anonymized data will be gathered and compared across the three wards. We have estimated that 90 (45+45) participants are required in order to meet our aims. In order to provide an answer as to whether this treatment is cost effective for the department by comparing total number of bed days, ward level of violence and wards cost of medication, we have calculated that we need a larger sample size of approximately 200 (100+100). We have implemented the broad consent at the Department of Acute Psychiatry and based on our experience, only 30-40 % of the patients choose to or are able to consent to research even when they are stable. We therefore expect that the intervention period will go on for approximately 6 months in order to achieve the number needed.

Due to the corona outbreak, the inclusion of patients for the AkuSleep study has been postponed indefinitely. The ward that was dedicated to the intervention has been transformed to a specialized unit treating psychiatric patients with either known COVID-19 or having symptoms of COVID-19. The study will start including patients when the Norwegian Health authorities have declared the outbreak to be under control and the ward is again offering standard treatment to patients with psychotic disorders.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to th he Acute Psychiatric Department at Oslo University who are able to consent

Exclusion Criteria:

* Patients not able to consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of sleep | 10 months
  Nursing staff report hours of sleep and number of awakening based on their observations which are recorded in the clinical record by night staff. All patients who receive treatment will be offered the opportunity to keep a sleeping diary for psycheducative purposes. The patients who are able to, will fill out the Insomnia Severity Index which is a brief instrument for assessment of sleep disturbances. In addition all patients, except those who cannot wear one for security reasons, will be offered an actigraph which provides the patient with a clear picture of their sleeping pattern. Relevant data from these actigraphs will be noted in the patients' clinical records.

SECONDARY OUTCOMES:
Psychotic symptoms | 10 months
  Current psychotic symptoms will be rated with the 6-item version of the Positive and Negative Syndrome Scale (PANSS).
Mania symptoms | 10 months
  Current manic symptoms will be rated using the Young Mania Rating Scale (YMRS).
Depressive symptoms | 10 months
  Depressive symptoms will be assessed with the Montgomery and Åsberg Depression Rating Scale (MADRS).
Psychosocial functioning | 10 months
  Psychosocial functioning in patients will be assessed with the Global Assessment of Functioning (GAF) scale, split version.
Brøset Violence Checklist (BVC) | 10 months
  BVC is a short-term violence prediction instrument assessing the six items confusion, irritability, boisterousness, verbal threats, physical threats and attacks on objects as either present of absent. The BVC is scored at every shift and at a scale ranging from 0-6 depending of the number of items present. Scores of 0 is considered low risk of imminent violent risk. A score of 1-2 predicts a moderate risk of violence and where preventive measures are advised and scores above 2 predict a high risk and preventive measures are necessary to secure safety.
Nursing category (PK-score) | 10 months
  Categories 1 and 2 describe patients that might be in need of some motivational support, but are aware of their condition and their needs and have the ability to take an active part in their own treatment. Global assessment of function scores (GAF) are typically in the above 45 range.Categories 3 and 4 describe patients with a clear need of nursing assistance. GAF scores are above 35. There is a need for consecutive risk assessments. The patients in these categories have a limited understanding of their condition and their need for treatment and limited ability to take part in planning of treatment. Patients in categories 3 and 4 are typically in need of hospital treatment. Categories 5 to 7 describe patients where there is an established to imminent risk of harm to self and/or others, where impulse control is failing and where the patient's ability to self-care is declining.
Disease severity | 10 months
  Number of days receiving involuntary treatment.
Number of days of stay. | 10 months
  Number of days that the patient is admitted before discharge.
Average bed days per ward. | 10 months
  Average number of bed days for each psychosis ward.
Aggressive events | 10 months
  Number of unwanted aggressive events as registered in clinical records and in the Hospital's reporting system (Achilles).
Medication | 10 months
  The current medication will be obtained through the medical records. Defined daily dosages (DDD) will calculated in accordance with the guidelines from the World Health Organization Collaborating Center for Drug Statistics Methodology (hhtp://www.whocc.no/atcdd). Total use of medication per ward.
Patient satisfaction | 10 months
  Upon discharge patients will be asked to fill out the Psychiatric Inpatient Questionnaire (PIPEQ) for rating their satisfaction with the treatment.

OTHER OUTCOMES:
Diagnosis | 10 months
  Diagnoses for description of demographics and adjustments in statistical analyses.
Age | 10 months
  Age for description of demographics and adjustment in statistical analyses.
Sex | 10 months
  Sex for description of demographics and adjustment in statistical analyses.
Disease duration | 10 months
  Disease duration for description of demographics and for adjustment in statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Dieset, MD/PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No